CLINICAL TRIAL: NCT00947895
Title: Relative Efficacy of Repeat Course of Intravenous methyLprednisolone and Intramuscular ACTH in the Treatment of Acute Relapse of Multiple Sclerosis After Sub Response to Initial Course of Intravenous Methylprednisolone (RECLAIM): a Single Center Pilot Study
Brief Title: Efficacy Study of Adrenocorticotropin Hormone to Treat Multiple Sclerosis (MS) Relapses After Sub-responding to an Initial 3 Day Course of Intravenous (IV) Methylprednisolone
Acronym: RECLAIM
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study reached halfway point in approximately one year time period and was halted to analyze data.
Sponsor: Neurologique Foundation, Inc. (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q1001
Record Dates: First submitted 2009-07-02; First posted 2009-07-28 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis
Keywords: ACTH; Acthar gel; adrenocorticotropin; methylprednisolone; solumedrol; MS; multiple; sclerosis; relapse; exacerbation; sub-responsive; IV
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis; Recurrence | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylprednisolone (Active Comparator): Intravenous (IV) methylprednisolone (Solumedrol) 1000 mg daily for 3 days.
  Interventions: Drug: Methylprednisolone; Other: IM placebo
- ACTH (Active Comparator): Intramuscular (IM) ACTH 80 mg/day for 5 days.
  Interventions: Drug: ACTH; Other: IV placebo

INTERVENTIONS:
Drug: Methylprednisolone — IV 1000 mg daily for 3 days
  Other Names: Solumedrol
  Arms: Methylprednisolone
Drug: ACTH — IM ACTH 80 mg/day for 5 days.
  Other Names: H.P. Acthar Gel; Repository corticotropin injection; Adrenocorticotropin hormone
  Arms: ACTH
Other: IV placebo — IV placebo (saline) daily for 3 days.
  Arms: ACTH
Other: IM placebo — IM placebo (saline) daily for 5 days.
  Arms: Methylprednisolone

SUMMARY:
The purpose of this study is to compare intramuscular (IM) ACTH (adrenocorticotropin hormone) and intravenous (IV) methylprednisolone (Solumedrol) for the treatment of an MS (Multiple Sclerosis) relapse (exacerbation) after sub-response to an initial 3 day course of IV methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

* male or female

  * females of childbearing potential must:

    * have negative pregnancy tests prior to entry into the Double-blind Treatment Phase
    * agree to use adequate contraception during the treatment.
  * females who are either post-menopausal for 12 months prior to randomization or surgically sterile (if documented), may be included without above requirements
* ≥ 18 years of age
* sign written informed consent prior to participating in the study (Appendix 1)
* willing and able to comply with trial requirements, including visit schedule and completion of scales
* diagnosis of multiple sclerosis by 2005 revised McDonald criteria (Appendix 3)
* an Expanded Disability Status Scale (EDSS) score of 0-6.0 inclusive
* currently taking a stable dose of an injectable MS disease modifying agent for the preceding 6 months or greater prior to the study-entry relapse
* in the opinion of their treating physician should undergo a 3 - 5 day course of IV methylprednisolone

Exclusion Criteria:

* a manifestation of MS other than relapsing
* initial IV MP greater than 14 days after from start of presenting relapse
* a history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome
* a known or 'new' diagnosis of diabetes mellitus (if screening blood glucose is suspicious for diabetes [≥126 mg/dL or ≥7 mmol/L if fasting; ≥200 mg/dL or 11.1 mmol/L if random testing] a patient should be further evaluated for diabetes mellitus)
* a contraindication to steroid therapy, e.g., peptic ulcer, psychotic states or severe hypertension
* sensitivity to proteins of porcine origin
* a known or 'new' diagnosis of severe depression as defined by a score greater than 30 on the Beck Depression Inventory (BDI)
* a known or 'new' diagnosis of hypothyroidism not adequately controlled with medication
* treatment with Natalizumab in the past 6 months
* active systemic bacterial, viral or fungal infections, or diagnosis of AIDS, Hepatitis B, Hepatitis C infection defined as a positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests, respectively
* have received total lymphoid irradiation or bone marrow transplantation
* have been treated with corticosteroids or adrenocorticotropic hormones (ACTH) within 1 month prior to Pre-Randomization Phase
* any medically unstable condition, as assessed by the primary treating physician
* any of the following neurologic/psychiatric disorders:

  * history of substance abuse (drug or alcohol) or any other factor (i.e., serious psychiatric condition) that may interfere with the subject's ability to cooperate and comply with the study procedures;
  * progressive neurological disorder, other than MS, which may affect participation in the study or require the use of medications not allowed by the protocol
* any of the following abnormal laboratory values:

  * serum creatinine greater than 1.7 mg/dL (150 μmol/L)
  * white blood cell (WBC) count <3,500/mm3 (<3.5 X 109 / L)
  * lymphocyte count <800/mm3 (<0.8 X 109 / L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Improvement in EDSS (Expanded Disability Status Scale) and Kurtzke Functional Scale (to assess individual disabilities). | 12 weeks

SECONDARY OUTCOMES:
Improvement in MSFC (Multiple Sclerosis Functional Composite)18 and its three individual components. | 12 weeks
Safety and tolerability of ACTH and MP in patients with an acute relapse of multiple sclerosis after sub-response to an initial course of intravenous methylprednisolone. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kantor, MD, Principal Investigator — Neurologique Foundation, Inc.
Locations (1):
- Neurologique Foundation, Inc., Ponte Vedra, Florida, United States

REFERENCES:
- See also: Study sponsor website — http://www.neurologique.org